CLINICAL TRIAL: NCT02446535
Title: REST/Collaborative Study Initiative With the Aim of Providing More Objective Information on Volume Status and Guiding Physicians in the Quest for DW
Brief Title: Probing the Dry Weight (DW) by Bioimpedance (BIA): Which is the Gold Standard Between Clinical DW and BIA DW?
Acronym: REST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Miulli General Hospital (Other)
Responsible Party: Principal Investigator, Carlo Basile, M.D., Scientific Director of the Division of Nephrology, Miulli General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MiulliGH
Record Dates: First submitted 2015-04-26; First posted 2015-05-18 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Uremia; Complication of Hemodialysis
MeSH Terms: conditions — Uremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BIA DW assessment (Experimental): All patients have undergone a Clinical DW assessment. Then, they undergo HD sessions in which BIA DW is determined reducing body weight (kg): when flattening of the BIA resistance occurs, the BIA DW is achieved and compared with the Clinical DW
  Interventions: Other: achievement of the DW by means of the BIA DW (RE.S.T.)

INTERVENTIONS:
Other: achievement of the DW by means of the BIA DW (RE.S.T.)

SUMMARY:
Background Very recently, a test aimed at assessing dry weight (DW) in hemodialysis (HD) patients has been developed, the "resistance stabilization test" (REST)

Aim of the study To verify if BIA-based DW (BIA DW) control is truly superior to current volume management in HD patients.

Protocol of the study DW determined with clinical methods (Clinical DW) is the gold standard by definition: Clinical DW is determined under strict clinical surveillance by the same attending physician. He will be helped by a clinical score of volume state about symptoms and signs of hypo- or hypervolemia. The physician is asked to adjust the DW of the candidates until their clinical score reaches zero before the BIA measurement. This Clinical DW will be compared with BIA DW, as obtained after performing REST

Phases of the study

The protocol study includes three sequential phases:

1. the Clinical DW is the gold standard by definition. Items of form B must be strictly applied until score = 0 is achieved;
2. The Clinical DW as indicated by the score = 0 becomes the target DW of the next standard HD session, in which BIA measurements are performed: R values are recorded continuously during the session.
3. REST is performed the following dialysis session. As per protocol, these dialysis sessions may be one or more than one, until flattening of the curve of the ratio R0/Rt (R0 is R at time 0 and Rt is R at a given time t during the HD session) of less than + 1% over 20 minutes in the presence of ongoing UF, is obtained.

Primary outcome

The primary outcome is the definition for each patient of the gold standard DW when comparing the Clinical and the BIA DW. Two are the possible scenarios:

1. the Clinical and the BIA DW will be very similar ( < + 0.5 kg). Therefore, a reciprocal validation of the two methods for that specific patient has been obtained;
2. the Clinical and the BIA DW are different ( > + 0.5 kg). If the BIA DW will be confirmed in the following six dialysis sessions, it means that the gold standard DW for that patient is the BIA DW.

DETAILED DESCRIPTION:
Background Probing the dry weight (DW) was largely dependent on clinical subjective estimates until recently. New bedside non-invasive tools have been developed with the aim of providing more objective information on volume status and guiding physicians in the quest for DW. Among them, bioimpedance (BIA) appears to be very promising in the achievement of this goal. Resistance (R) and capacitance of tissues are the two basic properties in BIA. However, although impedance is an electrical property of tissues that can be directly used in body composition analysis, it is commonly embedded in predictive equations that are derived by correlation with criterion measures of body compartments.

Very recently, a test aimed at assessing DW in hemodialysis (HD) patients has been developed, the "resistance stabilization test" (REST). It is based on the following four items:

1. one or more daily and/or alternate day HD sessions lasting 6 hours with ultrafiltration (UF) rate ≤ 0.5 kg/hour are planned;
2. BIA measurements are determined injecting 800 microAmpere at 50 kilohertz alternating sinusoidal current with a standard tetrapolar technique (BIA 101 Impedance Analyzer). Resistance (R) is recorded starting at the beginning of the HD session (R0) and then, continuously, until the end of the 6-hour session;
3. DW is defined as the weight achieved after flattening of the curve of the ratio R0/Rt (R0 is R at time 0 and Rt is R at a given time t during the HD session) of less than + 1% over 20 minutes in the presence of ongoing UF, indicating no further decline in extracellular volume;
4. if at the end of the 6-hour HD session R stabilization is not attained, a new 6-hour HD treatment with UF rate ≤ 0.5 kg/h is planned until a BIA DW (according to the item 3) is obtained.

Aim of the study A study group is being created (REST/Collaborative Study Initiative) with the aim of verifying if BIA-based DW (BIA DW) control is truly superior to current volume management in HD patients.

Protocol of the study DW determined with clinical methods (Clinical DW) is the gold standard by definition: Clinical DW is determined under strict clinical surveillance by the same attending physician. He will be helped by a clinical score of volume state about symptoms and signs of hypo- or hypervolemia. The physician is asked to adjust the DW of the candidates until their clinical score reaches zero after a given number of HD sessions before the BIA measurement. This Clinical DW will be compared with BIA DW, as obtained after performing REST;

Phases of the study

The protocol study includes three sequential phases:

1. as already mentioned, the Clinical DW is the gold standard by definition. Items of form B must be strictly applied. Form B must be filled in session after session, until score = 0, index of euvolemia, is achieved;
2. The Clinical DW as indicated by the score = 0 becomes the target DW of the next standard HD session, in which BIA measurements are performed: R values are recorded continuously during the session (Form C must be filled in).
3. REST is performed the following dialysis session (all the details have been given in the background section). As per protocol, these dialysis sessions may be one or more than one, until flattening of the curve of the ratio R0/Rt (R0 is R at time 0 and Rt is R at a given time t during the HD session) of less than + 1% over 20 minutes in the presence of ongoing UF, is obtained.

ELIGIBILITY:
Inclusion criteria:

1. patients older than 18 years
2. maintenance HD three times weekly.

Exclusion criteria:

1. dialysis vintage < 3 months
2. overt edema
3. liver cirrhosis
4. cardiac failure
5. serum albumin < 3 g/dl
6. pregnancy
7. metallic implants or a pacemaker
8. limb amputation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Bioimpedance (BIA) appears to be useful for the achievement of DW. Resistance (R, measured in Ohm) is a basic property of BIA. Postdialytic weight (kg) is measured with a bed scale. R and DW will be reported in the outcome measure data tables | up to 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology and dialysis unit Miulli General Hospital, Acquaviva delle Fonti, Bari, Italy